CLINICAL TRIAL: NCT04667052
Title: An Open-label, Randomized, Parallel Group Study to Assess the Relative Bioavailability of Two Different Subcutaneously-Administered JNJ-64304500 Formulations in Healthy Participants
Brief Title: A Study to Compare Two Different Subcutaneously-administered JNJ-64304500 Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108796; 64304500CRD1002 (Other: Janssen Research & Development, LLC); 2020-003559-14 (EudraCT Number)
Record Dates: First submitted 2020-12-09; First posted 2020-12-14 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ 64304500: Reference (Experimental): Participants (including individuals of Han Chinese background) will be randomized to receive a single subcutaneous dose of JNJ-64304500 reference formulation.
  Interventions: Drug: JNJ 64304500
- JNJ 64304500: Test (Experimental): Participants (including individuals of Han Chinese background) will be randomized to receive a single subcutaneous dose of JNJ-64304500 test formulation.
  Interventions: Drug: JNJ 64304500

INTERVENTIONS:
Drug: JNJ 64304500 — Participants will receive a single subcutaneous dose of JNJ-64304500 reference formulation.
  Arms: JNJ 64304500: Reference
Drug: JNJ 64304500 — Participants will receive a single subcutaneous dose of JNJ-64304500 test formulation.
  Arms: JNJ 64304500: Test

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of JNJ-64304500 after administration of two different formulations in healthy participants.

ELIGIBILITY:
Inclusion criteria:

* Male or non-childbearing potential female (according to their reproductive organs and functions assigned by chromosomal complement)
* For Han Chinese participants, they need to have resided outside of China for no more than 10 years and have parents and maternal and paternal grandparents who are of Han Chinese ethnicity
* Have a body weight in the range of 60 kilograms (kg) to 90 kg and within a body mass index range between 18 and 30 kilogram per square meters (kg/m^2), inclusive
* Healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) performed at screening.
* Healthy on the basis of clinical laboratory tests performed at screening.

Exclusion criteria:

* History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to) liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has a QT corrected according to Fridericia's formula (QTcF) interval greater than (>) 450 milliseconds (msec) for males, and >470 msec for females, has a complete left or right bundle branch block, or has a history or current evidence of additional risk factors for torsades de pointes (for example, heart failure, hypokalemia, family history of Long QT Syndrome) at screening and at predose (Day -1)
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Had major illness or surgery, (for example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from illness or surgery, or has surgery planned during the time the participant is expected to participate in the study or until Day 113 (Participants who had minor surgical procedures conducted under local anesthesia within 4 weeks before screening may participate)
* Plans to undergo non-major elective surgery within 4 weeks prior to study intervention administration through the end of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of JNJ-64304500 | Up to Day 113
  Cmax is the maximum observed serum concentration.
Area Under the Serum Concentration - Time Curve From Time Zero to Time Infinity (AUC [0-infinity]) of JNJ-64304500 | Up to Day 113
  AUC (0-infinity) is the area under the serum concentration-time curve from time zero to infinity time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the serum concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable concentration, and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 113
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are events between administration of study drug and up to Day 113 that are absent before treatment or that worsen relative to pre-treatment state.
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to Day 113
  Number of participants with clinically significant vital signs (temperature, pulse/heart rate, respiratory rate, and blood pressure: systolic and diastolic) will be reported.
Number of Participants with Clinically Significant Abnormalities in Physical Examinations | Up to Day 113
  Number of participants with clinically significant abnormalities in the physical examination (includes basic assessment of general appearance, respiratory and cardiovascular systems and the assessment of the skin at the administration area) will be reported.
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | Up to Day 113
  Number of participants with clinically significant abnormalities in laboratory assessments like serum chemistry, hematology, and urinalysis will be reported.
Number of Participants with Serum Antibodies to JNJ-64304500 | Up to Day 113
  Number of participants with serum antibodies to JNJ-64304500 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- WCCT Global, LLC, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency